CLINICAL TRIAL: NCT03301584
Title: Early Coordinated Rehabilitation in Acute Phase After Hip Fracture - a Model for Increased Patient Participation.
Brief Title: Early Coordinated Rehabilitation After Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Axel Linders Stiftelse (Unknown); SKLs' äldresatsning (Unknown); Local Research and Development Fund in Gothenburg and South Bohuslän (Unknown); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoU in Sweden 62221
Record Dates: First submitted 2017-09-22; First posted 2017-10-04 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Hip Fractures; Rehabilitation
Keywords: Hip fracture; ADL; patient participation; functional balance; physical performance
MeSH Terms: conditions — Hip Fractures; Patient Participation

STUDY DESIGN:
Intervention Model Description: A prospective, controlled, intervention study. Evaluation of a modified model of in-patient rehabilitation compared to standard care, with follow-up at 1 month post-discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced collaboration (Active Comparator): Enhanced OT and PT collaboration to promote patient participation. Goal setting using TLS-BasicADL protocol. Patients were encouraged to consider activities important to them to be able to perform at discharge. Adaption of goals throughout the hospital stay.
  Supporting patient self-efficacy: by challenging patients' fear of falling and encouraging progression of exercise.
  Training kit with instructions: To increase activity and encourage patients to take more responsibility for their training.
  Enhanced exercise with protocol: More intensive training of transfers, walking, balance and P-ADL was offered at least 3 times/day by OT and PT.
  Collaboration meetings: twice weekly interdisciplinary meetings plus daily OT and PT logistic meeting to schedule treatment.
  Interventions: Other: Enhanced collaboration to promote patient participation
- Usual Care Treatment (Active Comparator): Standard rehabilitation
  Interventions: Other: Usual Care treatment

INTERVENTIONS:
Other: Enhanced collaboration to promote patient participation — Enhanced OT and PT collaboration: to promote patient participation. Goal setting using TLS-BasicADL protocol. Patients were encouraged to consider activities important to them to be able to perform at discharge. Adaption of goals throughout the hospital stay.
  Supporting patient self-efficacy: by challenging patients' fear of falling and encouraging progression of exercise.
  Training kit with instructions: To increase activity and encourage patients to take more responsibility for their training.
  Enhanced exercise with protocol: More intensive training of transfers, walking, balance and P-ADL was offered at least 3 times/day by OT and PT.
  Collaboration meetings: twice weekly interdisciplinary meetings plus daily OT and PT logistic meeting to schedule treatment.
  Arms: Enhanced collaboration
Other: Usual Care treatment — The control group received standard rehabilitation from occupational therapists and physiotherapists (Monday to Friday), planned individually and gradually progressed for each patient. Mobilisation was initiated within 24 hours after surgery, 7 days a week. Patients were provided with a booklet with information about the fracture, operation method, exercise regime and assistive walking and ADL aid available.
  Arms: Usual Care Treatment

SUMMARY:
Background Studies have shown that patients with hip fracture treated in a Comprehensive Geriatric Care (CGC) unit report better results in comparison to orthopaedic care. Furthermore, involving patients in their healthcare by encouraging patient participation can result in better quality of care and improved outcomes. To our knowledge no study has been performed comparing rehabilitation programmes within a CGC unit during the acute phase after hip fracture with focus on improving patients' perceived participation and subsequent effect on patients' function.

Method A prospective, controlled, intervention performed in a Comprehensive Geriatric Care (CGC) unit and compared with standard CGC. A total of 126 patients with hip fracture were recruited who were prior to fracture; community dwelling, mobile indoors and independent in personal care. Intervention Group (IG): 63 patients, mean age 82.0 years and Control Group (CG): 63 patients mean age 80.5 years. Intervention: coordinated rehabilitation programme with early onset of patient participation and intensified occupational therapy and physiotherapy after hip fracture surgery. The primary outcome measure was self-reported patient participation at discharge. Secondary outcome measures were: TLS-BasicADL; Bergs Balance Scale (BBS); Falls Efficacy Scale FES(S); Short Physical Performance Battery (SPPB) and Timed Up and Go (TUG) at discharge and 1 month and ADL staircase for instrumental ADL at 1 month.

DETAILED DESCRIPTION:
At Sahlgrenska University Hospital patients with hip fracture are treated from admission to discharge in a CGC. To our knowledge no study has been performed within a CGC unit to compare rehabilitation programmes during the acute phase after hip fracture with focus on improving patients' perceived participation and the effect on patients' function.

The primary aim was therefore to evaluate a modified programme of coordinated inpatient rehabilitation during the acute phase after hip fracture surgery with focus was on patients' perceived participation. Secondary aims were to investigate effect on activities of daily living, functional balance and confidence and physical performance. A further aim was to investigate level of recovery at 1 month follow-up including risk for future falls.

Method Study design A prospective, controlled, intervention study. Evaluation of in-patient rehabilitation with follow-up at 1 month post-discharge.

Setting and Participants This study was performed in a CGC unit, at Sahlgrenska University Hospital in Gothenburg, Sweden comprising three wards, with a total of 78 beds. During September 2013 and May 2014, a convenience sample of 126 patients with hip fracture was recruited. Patients were admitted to one of the three wards depending on available beds. One ward was allocated as the intervention ward and the other two as controls.

Comprehensive Geriatric Care (CGC) All three geriatric wards follow a structured, systematic interdisciplinary geriatric care pathway for hip fracture patients, commencing at admission pre-operatively through to discharge. This follows a fast track approach including; assessment and management of the patient's somatic and mental health, physical function, ADL ability, social situation, early mobilisation/rehabilitation and early discharge planning. While orthopaedic surgeons are responsible for surgical fixation of the patients' fracture and routine examination of X-rays after the patient has been weight-bearing, patients are admitted to and cared for throughout their hospital stay by the interdisciplinary team on the geriatric ward.

Control:Usual Care Treatment The control group received standard rehabilitation from occupational therapists (OT) and physiotherapists (PT) (Monday to Friday), planned individually and gradually progressed for each patient. Mobilisation with weight-bearing of operated hip was initiated within 24 hours after surgery, seven days a week. Patients were provided with a booklet with information about the fracture, operation method, exercise regime and assistive walking and ADL aid available. Information was collected using TLS-BasicADL [26] regarding the patient's previous levels of physical function and ability to perform activities of daily living (ADL) and assessment of present ability performed as the patient was able. Patients received treatment by a PT on a daily basis (Monday to Friday) including mobilisation and progression of their exercise program, the number of times varied depending on patients' needs and staff resources. Interdisciplinary team meetings were held twice weekly to discuss progress and future planning. For those patients returning to own home, an OT prior to discharge, instructed them in the use of ADL aids, and assessed the need for aids in the home environment. All patients received both written and verbal information regarding prevention of falls prior to discharge.

Intervention

Psychological component:

Enhanced OT and PT collaboration: In addition to standard rehabilitation, focus was placed on promoting patient participation through closer collaboration between the OT and PT together with the patient. Patients were encouraged to take a more active part in and personal responsibility for their training and setting of rehabilitation goals. This involved, the OT and PT meeting the patient together within 24 hours postoperatively, they explained their roles in the inpatient rehabilitation process as facilitators to guide the patients in their recovery process while at the same time it was important that the patient felt involved and part of the team.

Goal setting using TLS-BasicADL: TLS-BasicADL protocol was used as in standard practice, however, an additional column for setting goals was added for the purpose of this study. Patients were encouraged, using the TLS-BasicADL protocol, to consider activities that were important to them to be able to perform at discharge. They were invited to answer the following question; "Which activities are important for you to achieve during your inpatient care?" The individual goals were followed up and adapted throughout the hospital stay using the TLS-BasicADL protocol.

Supporting patient self-efficacy: To strengthen patient's self-efficacy by challenging their fear of falling and encouraging patients' to progress their exercise. This was done under supervision of OT and PT with the aim that patients would gain confidence to take increased responsibility.

Physical component:

Training kit with instructions: To increase activity and encourage patients to take more responsibility for their training out with OT and PT treatment sessions, participants were provided with a training kit consisting of a sliding sheet and leg band to facilitate transfers in/out of the bed, a reaching aid, and stocking aid for training of ADL. Written and photographic instructions were included in the kit. All patients were given self-training exercises to perform daily to suit their level of dependence, adapted and intensified as the patient progressed.

Enhanced exercise with protocol: More intensive training of transfers, walking, balance and P-ADL was offered at least 3 times/day by OT and PT (Monday-Friday) from day 2 after surgery compared to control group. OT and PT filled in a training protocol showing when and how often patients received treatment. In addition the patients were encouraged to fill in an exercise diary.

Collaboration meetings: Over and above the twice weekly interdisciplinary meetings, the OT and PT met on a daily basis to plan daily training schedules to avoid collision. An additional meeting was held once a week, to further discuss routines concerning collaboration and treatment plans for individual patients. Patients were continually given feedback concerning their progress using TLS-BasicADL protocol.

Patients were asked daily about adverse reactions to treatment such as increased pain or fatigue, should this occur, events were documented in the patient records and treatment adapted as required.

Staffing levels and assessors The OT and PT staffing levels were similar on all three wards, with approximately 0.12 OT and PT per patient. Staff working on the two control wards were informed that the study was in progress, but no information was given regarding the content of the intervention, nor did they treat patients included in the intervention. The two OTs and three PTs who assessed the patients at discharge and one month were not blinded to the intervention but had no treatment association with the study patients.

Outcome Measures Demographic characteristics Pre-fracture baseline data were collected using a specifically designed study questionnaire covering social and living conditions, use of walking aids, frequency of outdoor walks with or without company, and level of social home service/informal help. Data concerning the fracture and other medical conditions were collected from medical records. At discharge, length of hospital stay and discharge destination were reported.

ELIGIBILITY:
Inclusion Criteria:

* presenting with acute hip fracture
* aged 65 or more
* able to speak and understand Swedish
* community dwelling pre-fracture
* independent walking indoors with or without walking aid and in personal care with exception of bathing/showering.

Exclusion Criteria:

* severe drug or alcohol abuse
* mental illness
* documented cognitive impairment ≤ 8 according to the Short Portable Mental Status Questionnaire (SPMSQ)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Self-rated degree of patient participation in rehabilitation | At discharge from in-patienten rehabilitation, on average 14 days
  Patients answered 4 questions, specifically formulated for this study, regarding perceived level of participation in; their rehabilitation; working together with OT and PT in goal-setting; personal responsibility for their training, and making decisions regarding care and treatment as much as they liked. The questions were answered using a four level scale; very high degree, moderate degree, small degree or not at all.

SECONDARY OUTCOMES:
Traffic Light System - BasicADL (TLS-BasicADL) | At discharge from in-patient rehabilitation, on average 14 days and 1 month follow-up
  TLS-BasicADL highlights the patient's level of independence in basic ADL, comprising of 15 different activities; 6 items showing ability to transfer and walk indoors, 7 P-ADL items and 2 additional items; negotiating stairs and walking outdoors. Three colour-coded markers indicate level of dependence; green=independent, yellow=supervision and red=dependent on physical help of others. TLS-BasicADL does not form a composite score but shows through the colour-coding, level of dependence with regard to the patient's; 1) previous ability and assistive aids prior to admission to hospital, 2) present ability and assistive aids used and 3) goals which the patient aims to achieve during inpatient treatment. As the patient's ability to perform activities changes during in-patient rehabilitation, the colour-coded markers are changed correspondingly.
ADL Staircase | At 1 month follow-up
  Ability to perform instrumental activities of daily living was assessed using IADL items of the ADL-staircase.
  The ADL staircase is an expansion of Katz ADL Index of personal activities of daily living, with the addition of four I-ADL items; cooking, shopping, cleaning, and transportation. The ADL staircase uses only two levels; dependent or independent and can be administered through interview and/or observation. The ADL-staircase has shown good validity and reliability, and is considered a stable and clinically relevant when used in studied of older people.
Bergs Balance Scale (BBS) | At discharge from in-patient rehabilitation, on average 14 days and 1 month follow-up
  To measure functional balance and fall risk. BBS assesses 14 activities of varying difficulty with a scoring range from 0-4 (0 unable to perform to 4 able to perform completely). The item scores are summed giving a score of 0-56, with 56 showing indicating normal functional balance. BBS has shown excellent test-retest reliability and validity. To determine clinical significance, minimal detectable change (MDC) scores described by Donoghue & Stokes were used, ranging from 4-7 points depending on baseline score. To discriminate those at risk for falls, a cut-off score of 47 was defined.
Falls Efficacy Scale (FES-S) | At discharge from in-patient rehabilitation, on average 14 days and 1 month follow-up
  Balance confidence was measured using the Swedish version of the Falls Efficacy Scale (FES-S). This version is modified from the original 10-degree scale (1-10) where 1 represents 'very confident, no fear of falling' and 10 'not confident at all, very afraid of falling', into an 11-degree scale (0-10) with a reversed answering alternative (0 not confident at all and 10 totally confident). For the purpose of this study the aspect of confidence rather than fear has been assessed. FES-S includes 13 items, comprising three parts, six items measuring self-care, one item stair walking, and six items instrumental activities. The maximum score is 130. Test-retest reliability of the Swedish version of the scale was found to be acceptable by Hellstrom et al.
Short Physical Performance Battery (SPPB) | At discharge from in-patient rehabilitation, on average 14 days and 1 month follow-up
  Short Physical Performance Battery (SPPB) consists of three components: standing balance, walking speed - timed 4 m walk, and ability to rise from chair. The sum of the three components comprises the final SPPB score with a possible range from 0 to 12 (12 indicating the highest degree of lower extremity functioning). According to Perera et al a small meaningful change is 0.5 and a substantial meaningful change 1.0 point respectively. For analysis of risk for falls a score of ≤ 6 is associated with a higher fall rate.
Timed Up and Go (TUG) | At discharge from in-patient rehabilitation, on average 14 days and 1 month follow-up
  The Timed Up and Go (TUG) test measures ability to perform basic everyday movements. TUG assesses total time for standing up from a standard chair, walking 3m, turning 180 degrees, returning and sitting down. According to recommendations by Podsiadlo and Richardson, TUG was performed twice in each test session, one trial and one timed performance, with a brief seated rest in between. The participants were instructed to walk at a comfortable, safe speed. TUG has good inter-rater and intra-rater reliability and is a reliable and valid measure of functional mobility. A TUG score >24 seconds at discharge, was used for analysis of risk for falls, which is a predictor for falls at 6 months in hip fracture patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Zidén, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Mölndal Hospital, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- [Derived] Asplin G, Carlsson G, Ziden L, Kjellby-Wendt G. Early coordinated rehabilitation in acute phase after hip fracture - a model for increased patient participation. BMC Geriatr. 2017 Oct 17;17(1):240. doi: 10.1186/s12877-017-0640-z. PMID 29041916